**Trial Title:** STENT <u>RETRIEVE</u>R THROMBECTOMY FOR THROMBUS BURDEN REDUCTION IN PATIENTS WITH <u>A</u>CUTE <u>M</u>YOCARDIAL <u>I</u>NFARCTION – RETRIEVE – AMI study

Short title: RETRIEVE-AMI

Ethics Ref: 21/SC/0220

IRAS Project ID: 294665

Date and Version No: 22/04/2024 v4.0

Chief Investigator: Dr Giovanni Luigi De Maria

Department of Cardiology, John Radcliffe Hospital

Investigators: Prof Adrian P Banning

Department of Cardiology, John Radcliffe Hospital

Prof Keith M. Channon

Department of Cardiology, John Radcliffe Hospital

Dr Rafail A. Kotronias

Department of Cardiology, John Radcliffe Hospital

Dr Jeremy P. Langrish

Department of Cardiology, John Radcliffe Hospital

Dr Mohammad Alkhalil

The Newcastle upon Tyne Hospitals NHS Foundation Trust

**Sponsor:** Oxford University Hospitals NHS Foundation Trust

Research and Development Department

Joint Research Office

Oxford University Hospitals NHS Foundation Trust

Second Floor, OUH Cowley Unipart House Business Centre

Garsington Road Oxford OX4 2PG

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


Funder: Medtronic and Terumo Inc

**Chief Investigator Signature:** 

Labring Bannje Statistician Signature:

# **Confidentiality Statement**

This document contains confidential information that must not be disclosed to anyone other than the Sponsor, the Investigator Team, HRA, host organisations, and members of the Research Ethics Committee and Regulatory Authorities unless authorised to do so.

# 1. Table of Contents

| 2. KEY TI | EY TRIAL CONTACTS6 | |
|---|---|---|
| 3. Lay Su | Summary | |
| 4. SYNOI | SYNOPSIS8 | |
| 5. ABBRI | EVIATIONS | 9 |
| 6. BACKO | GROUND AND RATIONALE | 10 |
| 7. НҮРО | THESIS | 12 |
| 8. OBJEC | TIVES AND OUTCOME MEASURES | 12 |
| 9. TRIAL | DESIGN | 13 |
| | RTICIPANT IDENTIFICATION | |
| 10.1. | Trial Participants | |
| 10.2. | Inclusion Criteria | 15 |
| 10.3. | Exclusion Criteria | 15 |
| 11. TRIA | AL PROCEDURES | 17 |
| 11.1. | Informed Consent | 17 |
| 11.2. | Discontinuation/Withdrawal of Participants from Trial Treatment | 20 |
| 11.3. | Recruitment | |
| 11.4. | Randomisation | 21 |
| 11.5. | Blinding and code-breaking | 23 |
| 11.6. | Study timeline | 23 |
| 11.7. | Trial Assessments | 25 |
| 11.7.1. | Data Collection, Patient Reported Outcomes and Clinical Outcomes <u>Error! Bookmark I</u> | |
| 11.7.2.<br>11.7.3. | Optical Coherence Tomography<br>Angiography-derived coronary physiology | |
| 11.7.3. | Extracted Thrombus Imaging | |
| 11.7.5. | Electrocardiography (ECG) | |
| 11.8. | Subsequent telephone follow-ups | |
| 11.9. | Definition of End of Trial | 26 |
| 12. IDEI | NTIFICATION & DESCRIPTION OF THE INVESTIGATIONAL DEVICE & COMPAR | RATORS28 |
| 12.1. | Investigational Device & Comparators | 28 |
| 12.1.1. | Standalone PCI (Arm 1) | 28 |
| 12.1.2. | Aspiration thrombectomy and PCI (Arm 2) | 28 |
| 12.1.3. | Investigational arm (Arm 3) | 28 |
| 12.1.4. | Masking (blinding) | |
| 12.1.5. | Storage of investigational devices | 29 |
| 12.2. | Retriever thrombectomy safety | |

Deleted: 25

Clinical Trial Protocol Template version 15.0


 $\hbox{@ Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019}\\$ 

| | 12.3. | Other Interventions | 31 |
|---|---|---|---|
| 1 | 3. SAF | ETY REPORTING | 32 |
| | 13.1. | Definitions | 32 |
| | 13.2. | Causality | 35 |
| | 13.3. | Procedures for Recording Adverse Events | 36 |
| | 13.4. | Reporting Procedures for Serious Adverse Events | 36 |
| | 13.5. | Expectedness | 37 |
| | 13.6. | Trial cessation rules | 37 |
| | 13.7. | Safety Monitoring Committee – Trial Safety Group (TSG) | 37 |
| | 13.8. | Safety of stent-retriever thrombectomy | 38 |
| | 13.9. | Safety of intravascular imaging | 38 |
| 1 | 4. STA | TISTICS | 39 |
| | 14.1. | Number of participants | 39 |
| | 14.2. | Analysis of Endpoints | 39 |
| | 14.3. | Interim Safety Analysis | 40 |
| 1 | 5. DA1 | TA MANAGEMENT | 41 |
| | 15.1. | Source Data | 41 |
| | 15.2. | Data recording and Record Keeping | 41 |
| | 15.3. | Access to Data | 42 |
| | 15.4. | Approval to share imaging data with third parties | 42 |
| 1 | 6. QU | ALITY ASSURANCE PROCEDURES | 44 |
| | 16.1. | Risk assessment | 44 |
| | 16.2. | Monitoring | 44 |
| 1 | 7. PRC | DTOCOL DEVIATIONS | 45 |
| 1 | 8. SER | IOUS BREACHES | 45 |
| 1 | 9. ETH | IICAL AND REGULATORY CONSIDERATIONS | 46 |
| | 19.1. | Declaration of Helsinki | 46 |
| | 19.2. | Guidelines for Good Clinical Practice | 46 |
| | 19.3. | Medical Device Regulations | 46 |
| | 19.4. | Approvals | 46 |
| | 19.5. | Specific Ethical Considerations for participants in emergency situations | 47 |
| | 19.6. | Possible risks/discomfort to participants | 47 |

| 19 | 9.7. | Collaboration and Partnership with Commercial Companies & Third parties | . 48 |
|---|---|---|---|
| 19 | 9.8. | Feasibility | . 49 |
| 19 | 9.9. | Reporting | . 49 |
| 19 | 9.10. | Participant Confidentiality | . 49 |
| 20. | FIN | ANCE AND INSURANCE | .49 |
| 20 | 0.1. | Funding | . 49 |
| 20 | 0.2. | Insurance | . 50 |
| 21. | PUL | BLICATION POLICY | .50 |
| 22. | DE | /ELOPMENT OF A NEW PRODUCT/ PROCESS OR THE GENERATION OF INTELLECTUA | 4 <i>L</i> |
| PRC | PERTY | / | .50 |
| 23. | REF | ERENCES | .51 |
| 24. | API | PENDIX A: Trial flow chart | .54 |
| 25. | API | PENDIX B: Vessel reference diameters for device sizing | . 55 |
| 26. | | PENDIX C: Schematic diagram of device operation | |
| 27. | | PENDIX D: Amendment history | |
| <i>-/</i> . | AFF | - LIVDIA D. AIIICIIUIIICIII IIISIUI Y | |

# 2. KEY TRIAL CONTACTS

| . RET TRIAL CONTACTS | · |
|----------------------|--------------------------------------------------|
| Chief Investigator | Dr Giovanni Luigi De Maria |
| | Department of Cardiology |
| | John Radcliffe Hospital |
| | Headington, Oxford, OX3 9DU |
| | GiovanniLuigi.DeMaria@ouh.nhs.uk |
| | Tel: 07490707811 |
| Sponsor | Oxford University Hospitals NHS Foundation Trust |
| | Research and Development Department |
| | Joint Research Office |
| | Oxford University Hospitals NHS Foundation Trust |
| | Second Floor, OUH Cowley |
| | Unipart House Business Centre |
| | Garsington Road |
| | Oxford OX4 2PG |
| | ouh.sponsorship@ouh.nhs.uk |
| Funder(s) | Medtronic and Terumo Inc |
| Clinical Trials Unit | Net applicable |
| Clinical Trials Unit | Not applicable |
| Statistician | Dr Abhirup Banerjee |
| | Division of Cardiovascular Medicine |
| | Radcliffe Department of Medicine |
| | University of Oxford |
| | abhirup.banerjee@cardiov.ox.ac.uk |
| | Tel: +44 7448807087 |

3. Lay Summary

Heart attacks are caused by the sudden formation of a clot inside a diseased coronary artery which

reduces blood flow beyond the blockage site. During conventional treatment of the blockage with what is

known as a stent; a stainless-steel tube that keeps the artery open, the clot that has formed is disrupted

and is pushed further down leading to damage in smaller blood vessels supplying the heart muscle. This

additional damage can lead to long-term heart muscle damage influencing recovery and wellbeing. The

original concept that was tested to prevent this 'clot shower' was that of a suction device to withdraw the

clot before stenting. However, this approach has not translated to patient benefit.

Amongst the reasons put forward for the inefficacy of the suction device was that it does not remove

the entire clot as it does not interact with it. A new device that physically interacts with the clot and traps

it before pulling it out - the stent retriever - is now routinely used in stroke therapy to remove clots in the

arteries supplying the brain. This device has been successfully used as a last resort to remove clots in a

small number of heart attacks. We hypothesize that stent retriever therapy will be more effective in clot

removal than the current standard of care; suction or stenting. To study this, we propose the RETRIEVE-

AMI randomised controlled trial.

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


## 4. SYNOPSIS

| 4. SYNOPSIS | | | |
|---|---|---|---|
| Trial Title | STENT <u><b>RETRIEVE</b></u> R THROMBECTOMY FOR THROMBUS BURDEN REDUCTION IN PATIENTS WITH <b>A</b> CUTE <b>M</b> YOCARDIAL INFARCTION | | |
| Internal ref. no. (or short title) | RETRIEVE – AMI study | | |
| Trial registration | NCT05307965 | | |
| Sponsor | Oxford Univ | ersity Hospitals NHS Foundation Tru | ust |
| Funder | | Medtronic & Terumo Inc | |
| Clinical Phase | | Device Pilot | |
| Trial Design | R | andomised controlled trial | |
| Trial Participants | ST elevat | cion Myocardial Infarction Patients | |
| Sample Size | | n=81 | |
| Planned Trial Period | | Start Date: 01/03/2022<br>End Date: 30/09/2025 | |
| Planned Recruitment period | | 36 months | |
| 1 | Objectives | Outcome Measures | Timepoint(s) |
| Primary | Efficacy of thrombus burden reduction | Thrombus volume (mm³)<br>(OCT assessment) | Pre-stent |
| | Cofety of vetries on | Angiography-/OCT-defined<br>device related target vessel<br>complications, device | Pre-stent |
| Co-primary | Safety of retriever thrombectomy | deficiency Rate of major adverse cardiac and cerebrovascular events (MACCE) | In hospital<br>30 days<br>6 months |
| | Efficacy of thrombus burden reduction | Thrombus area, flow area (mm²) (OCT assessment) | Pre-stent |
| Secondary | Efficacy of<br>thromboatheroma<br>reduction | Thromboatheroma area, flow area (mm²) (OCT assessment) | Post-stent |
| | Efficacy of stent implantation | Stent expansion & apposition (OCT assessment) | Post-stent |
| | Angiographic success rate | TIMI flow, Myocardial Blush<br>Grade, Angiography derived<br>coronary physiology indices | Post-stent |
| Intervention(s) • Other intervention(s) | Percutaneous coronary intervention with adjunctive use of stent retriever thrombectomy | | |
| Comparator | | ry Intervention alone or Percutaneo<br>rith adjunctive aspiration thrombed | • |

# 5. ABBREVIATIONS

| AE | Adverse event |
|---|---|
| ADE | Adverse device effect |
| CI | Chief Investigator |
| CRF | Case Report Form |
| СТА | Clinical Trials Authorisation |
| CTRG | Clinical Trials and Research Governance |
| GCP | Good Clinical Practice |
| GP | General Practitioner |
| HRA | Health Research Authority |
| ICH | International Conference on Harmonisation |
| IRB | Independent Review Board |
| MACCE | Major adverse cardiac and cerebrovascular event |
| MHRA | Medicines and Healthcare products Regulatory Agency |
| NHS | National Health Service |
| RES | Research Ethics Service |
| ОСТ | Optical coherence tomography |
| OXTREC | Oxford Tropical Research Ethics Committee |
| PCI | Percutaneous coronary intervention |
| pPCI | Primary percutaneous coronary intervention |
| PI | Principal Investigator |
| PIL | Participant/ Patient Information Leaflet |
| R&D | NHS Trust R&D Department |
| REC | Research Ethics Committee |
| RMP | Registered Medical Practitioner |
| SAE | Serious Adverse Event |
| SADE | Serious Adverse Defice Effect |
| SOP | Standard Operating Procedure |
| TIMI | Thrombolysis in myocardial infarction |
| TMF | Trial Master File |
| TSG | Oxford University Hospitals NHS Foundation Trust Trials Safety Group |

#### 6. BACKGROUND AND RATIONALE

Ischaemic heart disease remains the leading cause of death across the globe despite sustained reductions in mortality rates.1 However, cardiovascular morbidity following myocardial infarction remains a significant burden to healthcare systems. Our attempts during the last decade have thus shifted towards reperfusion therapies that reduce the extent of the myocardial infarction.<sup>2</sup>

Amongst the proposed adjuncts to angioplasty, aspiration thrombectomy has been proposed as a simple method of removing the in-situ clot prior to stent deployment. Aspiration thrombectomy was thought to reduce distal embolisation of athero/thrombotic debris, limiting the ensuing microvascular dysfunction and final infarct size.  $^{3,4}$  Early randomised controlled trials of aspiration thrombectomy supported its routine clinical use,<sup>5</sup> but contemporary trials suggest no effect on mortality and a signal of increased stroke. 6.7 Amongst the reasons put forward to explain the lack of benefit of aspiration thrombectomy is its inefficacy in removing thrombi.8 Indeed, the optical coherence tomography (OCT) sub-study of TOTAL suggested that there was no difference in pre-PCI thrombus volume in lesions treated with aspiration thrombectomy versus PCI alone.9

One of the reasons why thrombus-aspiration catheters failed to remove thrombotic debris in STEMI can be related to the inability of the devices to actually interact with the clot. In the coronary artery the clot develops on top of an ulcerated/ruptured plaque, meaning that the bulk of the clot is often in an eccentric position, eventually protruding towards the centre of the lumen. An additional element that must be taken into account is the disproportion between the vessel lumen-cross-section-area (which can potentially be filled with thrombus) and the aspiration-opening area at tip of the aspiration catheter. If an average size coronary artery (diameter: 3.0 - 3.5 mm) is considered, the vessel lumen-cross-section-area can range from 7.06 to 9.61 mm<sup>2</sup>. Since the aspiration-opening area at tip of the aspiration catheter is on average 0.9-1.0 mm<sup>2</sup>, that means that the thrombectomy device technically covers (on average) from 9.4 to 14.2% of the vessel lumen-cross-section-area. In a larger caliber vessel (for example large ectatic right coronary arteries) this ratio becomes even more unfavourable. As the caliber of the vessel increases, its "theoretical" ability to contain large thrombus-burden increases proportionally, meaning that Clinical Trial Protocol Template version 15.0 CONFIDENTIAL © Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


paradoxically the currently available aspiration devices become less effective in those cases when they

would be required to work at their best.

Another element to account for poor performance of the current aspiration-catheters is the "guidewire

bias effect". This is a direct consequence of 1) the coronary arteries not being straight tubes, but having

bends and curves and 2) of the thrombectomy-catheter sliding over an angioplasty-guidewire during the

procedure. In a curved tube, like the coronary artery, the position of the wire can actually bias the

aspiration device away from the clot. The "guidewire bias effect" can be minimally influenced by the

operator. For this reason a clot-removal device that could interact with the whole vessel-lumen cross

section area (and thus with the whole clot) and whose mode action is not affected by coronary artery

caliber and by "guidewire bias effect" would be desirable and likely to be more effective in removing

thrombus in STEMI patients.

Stent-retriever thrombectomy technology has this property and not surprisingly it has revolutionised the

 $treatment\ of\ acute\ is chaemic\ stroke\ improving\ recanalization\ rates\ and\ clinical\ outcomes\ significantly. ^{10,11}$ 

Stent-retriever technology has been proved to be safe with low rates of vascular perforations (~2.1%) and

iatrogenic dissection (1.7%-3.5%) in acute ischaemic stroke treatment.  $^{10\text{-}14}$ 

Isolated case reports of successful bailout stent-retriever thrombectomy in ST elevation myocardial

infarction (STEMI) patients attest to the feasibility of a stent-retriever thrombectomy approach in

 ${\sf STEMI.}^{15,16} \ \ {\sf However} \ \ {\sf whether} \ \ {\sf a} \ \ {\sf stent-retriever} \ \ {\sf strategy} \ \ {\sf is} \ \ {\sf more} \ \ {\sf effective} \ \ {\sf that} \ \ {\sf conventional} \ \ {\sf thrombus}$ 

aspiration in STEMI has to be proved. Recently, stent retriever thrombectomy with the NeVa (Vesalio)

device was evaluated in STEMI patients with large thrombus burden. 17

We set out to study the efficacy and safety of retriever thrombectomy in a carefully selected cohort of

patients with ST elevation myocardial infarction and compare it with current standard of care; standalone

PCI or PCI with adjunctive thrombus aspiration. We expect that stent retriever thrombectomy will more

 $effectively\ reduce\ the\ thrombotic\ burden\ when\ compared\ to\ the\ current\ standard\ of\ care\ (e.g.\ standalone)$ 

PCI and/or PCI with adjunctive aspiration thrombectomy).

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


## 7. HYPOTHESIS

We hypothesize that stent retriever thrombectomy will be more efficacious than aspiration or mechanical thrombectomy in thrombus burden reduction as assessed by OCT derived pre-stent thrombus volume (mm³).

# 8. OBJECTIVES AND OUTCOME MEASURES

| Objectives | Outcome Measures | Timepoint(s) of evaluation of this outcome measure (if applicable) |
|---|---|---|
| Primary Objectives | | |
| Efficacy of thrombus burden reduction | Thrombus volume (mm³) (OCT assessment) | Pre-stent |
| | Angiography-/OCT-defined device | Pre-stent |
| Safety of retriever thrombectomy | related target vessel complications, device deficiency | In hospital |
| | <ul> <li>Rate of major adverse cardiac and<br/>cerebrovascular events (MACCE)</li> </ul> | 30 days |
| | | 6 months |
| Secondary Objectives | | |
| Efficacy of thrombus burden reduction | Thrombus area, flow area (mm²) (OCT assessment) | Pre-stent |
| Efficacy of thromboatheroma reduction | Thromboatheroma area, flow area (mm²) (OCT assessment) | Post-stent |
| Efficacy of stent implantation | Stent expansion & apposition (OCT assessment) | Post-stent |
| Angiographic success rate | TIMI flow, Myocardial Blush Grade,<br>Angiography derived coronary<br>physiology indices | Post-stent |

9. TRIAL DESIGN

RETRIEVE AMI is an investigator-initiated, multi-centre, exploratory three arms, randomised controlled

trial. Patients over the age of 18 admitted for primary PCI (pPCI) for ST elevation myocardial infarction and

meeting the inclusion criteria laid out in section 10.2 will be 1:1:1 randomised to receive either standalone

PCI (Arm 1), thrombus aspiration + PCI (Arm 2) or retriever thrombectomy + PCI (Arm 3). Recruitment is

expected to last for 18 months with the study finishing when the last follow-up of the last recruited patient

is completed and all data is entered into the study. Each participant is expected to remain in the study for

6 months during which one telephone follow-up at 6 months will be arranged. (Figure 1, Appendix A)

The RETRIEVE AMI will enrol specifically patients with

- evidence of large thrombus burden on coronary angiography

- with culprit lesion located in a relatively large caliber (diameter > 3.0 mm) coronary artery

By only including a large caliber vessel, the retriever-stent will be tested in a setting where the currently

available technology is perceived to be suboptimal as described in section 6. Our decision to expand

recruitment to the left coronary system was driven by our experience with the device in this trial as well

as from published reports of the systematic evaluation of the NeVa (Vesalio) stent retriever device. Indeed,

the authors have shown that thrombectomy is safe in both the left and right coronary artery systems. 17

Procedurally, we are reducing the risk of a major interaction of the device by placing a coronary guidewire

alongside the stent retriever allowing us to retain safe control of the vessel whilst the clot is retrieved.

Clinical Trial Protocol Template version 15.0




Figure 1: Trial flow chart

#### 10. PARTICIPANT IDENTIFICATION

#### 10.1. **Trial Participants**

Patients over 18 years of age having pPCI for ST elevation myocardial infarction and meeting the inclusion criteria as listed below will be randomised to either retriever thrombectomy + PCI, or thrombus aspiration + PCI, or standalone PCI.

#### 10.2. **Inclusion Criteria**

- Male or Female, aged 18-90 years.
- pPCI patient with ST elevation myocardial infarction.
- Angiographic criteria:
  - ♦ TIMI 0/1 flow at presentation
  - ♦ Angiographic thrombus score ≥ 4
  - $\Diamond$  Vessel diameter at site of occlusion  $\geq$  3.0 mm (measured by quantitative coronary angiography)

#### 10.3. **Exclusion Criteria**

The participant may not enter the trial if ANY of the following apply:

- Female participant who is pregnant or lactating
- Participant with known hypersensitivity to nickel-titanium
- Unconscious at presentation
- Late presenter (pain to wire time > 12 h)
- Class Killip III/IV and/or profound bradycardia (HR < 40 bpm)
- Known history of kidney failure
- Ostial occlusion

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


| Date and version | No:22/04/2024 v4 | n |
|------------------|-------------------|---|
| Date and version | NO:22/U4/2U24 V4. | u |

- Highly tortuous vessel\*
- Highly calcified vessel
- Suspected (angiographically) spontaneous coronary artery dissection
- Stent thrombosis
- Previous stent implanted proximal to the occlusion site
- Previous CABG
- Previous STEMI/TIA/Stroke
- Known anaemia (Hb <9).

Clinical Trial Protocol Template version 15.0


<sup>\*</sup>A highly tortuous vessel is defined by the presence of  $\geq$ 3 consecutive curvatures of 90° to 180° measured at enddiastole in a major epicardial coronary artery  $\geq$ 2 mm in diameter.\(^{18} In our protocol tortuosity will lead to a participant's exclusion if it is affecting the vessel at the target lesion or proximal to it.

#### 11. TRIAL PROCEDURES

#### 11.1. Informed Consent

Informed consent will be obtained, with the recruitment approach to the patient, as described below.

### 11.1.1. Waiver request for patients having emergency angioplasty procedure

The clinical treatment of these patients is in the emergency context and delays to treatment are detrimental. It is necessary to administer prompt emergency treatment and it is not always possible to identify and approach a Consultee beforehand. Thus we would seek a waiver, as described in Section 32(9) of the Mental Capacity Act, since

- a) the treatment needs to be given urgently,
- b) it is necessary to take the action for the purpose of the research urgently,

but

c) it is not reasonably practicable to consult prior to enrolling the patient.

In this situation the Mental Capacity Act allows the participant to be enrolled with an agreement of a registered medical practitioner (RMP) not involved in the research or in accordance with a procedure agreed with the appropriate body (i.e. REC). Since this is only applicable for the duration of the emergency we will seek written informed consent as soon as reasonably practicable (see diagram and Section 11.1.1.2 below). This process includes an important role for a healthcare professional as a type of patient "advocate". This is discussed in section 11.1.1.2 below. We also seek approval from the REC for the waiver procedure.

# 11.1.1.1. Verbal assent

Because of the urgency of the situation it is not feasible to obtain fully informed written consent. Fully informed consent requires that the potential participant have time to read and reflect on a patient information sheet which in this context is clinically inadvisable. We therefore propose to obtain verbal assent so as to optimize the amount of appropriate information conveyed to potential participants

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


acutely and minimize the clinical risks involved with substantial delay. The research study will be

discussed verbally with the patient and the risks and benefits explained.

In detail the patient at the time of verbal assent process will be informed that the particular pattern of

heart attack they are having would be suitable for recruitment in our research trial which investigates a

new device to remove the blood clot that is causing the heart attack. We will explain that as part of the

trial they will receive either standard of care procedures or the investigational device. We will also briefly

mention that we will be obtaining some extra pictures from within the arteries, a sample of the clot and

measurements of flow and resistance in the small net of capillaries feeding the heart.

Participants will be reminded that they have the right to withdraw from the study at any stage and that

this will not affect their treatment or human rights. The research and clinical team have extensive

experience of patient assent, and the role of a Patient Advocate (see below), through the recruitment of

approximately 500 participants undergoing emergency PCI for STEMI in the OxAMI [Ethics Ref

11/SC0397] and OxAMI PICSO [Ethics Ref 15/SC0167] studies. Newcastle upon Tyne Hospitals NHS

Foundation Trust is a participating site to the OxAMI Study.

Only conscious patients, able to provide verbal assent will be enrolled in the study.

11.1.1.2. Patient Advocate

Because of the urgency of the situation it is not feasible to obtain written informed consent from the

patient prior to enrolment, so an RMP or patient "advocate" will be identified to act in accordance with

section 32(9). The Patient Advocate will act as witness and documenter of the verbal assent process for

all conscious potential participants and/or overseer of the waiver process as a whole. This RMP will be

present at the time of emergency treatment, but is not part of the research team. The Advocate will

ensure that the verbal assent process is undertaken, that the patient does not object (i.e. the patient

"assents" rather than "dissents"), and that the researcher has taken practical steps to explain the study,

risks and benefits, within the context of the emergency clinical situation, and in accordance with the

clinical status of the patient. The Advocate in this situation will be a healthcare professional such as a

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


Commented [GS(O1]: I don't think this is needed here?

Commented [RK2R1]: It is as the assent relies on OxAMI

specialist nurse. Assessment of patients in this context is within their professional capacity and the role here will be to witness verbal assent.

Most of the nursing staff at the Oxford Heart Centre has already attended a series of seminars to make them aware of their specific roles and responsibilities in this situation, and they have acted as patients' advocates through the recruitment of approximately 500 participants undergoing emergency PCI for STEMI in the ongoing OxAMI and OxAMI PICSO studies. The seminars have been directed by an ethicist who is not directly involved with the research project. We will continue to provide this training and draw on the extensive experience of the members of the clinical team currently acting as a Patient Advocate. Staff training at the Newcastle upon Tyne University Hospitals NHS Foundation Trust is ongoing.



## 11.1.1.3. Post-emergency phase

Once the emergency phase is over and treatment has been delivered, we will seek full written informed consent as soon as practical. For most patients this means within 12 hours of admission. This consent will be a two parts process:

a) We will seek consent to allow use of data already acquired during the emergency phase

Clinical Trial Protocol Template version 15.0


 $^{\circ}$  Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019 

b) We will seek consent for ongoing participation in the study.

Written Informed Consent will be obtained by means of participant dated signature and dated signature of the person who presented and obtained the Informed Consent. The person who obtained the consent must be suitably qualified and experienced, and have been authorised to do so by the Chief/Principal Investigator. A copy of the signed Informed Consent will be given to the participant and another copy will. Be filed in their medical records. The original signed form will be retained at the trial

site.

If the participant elects to withdraw from the study at this point then we will present them with three withdrawal options as outlined in section 11.2.1.

If a patient is unable to provide informed consent at this stage due to deterioration in clinical condition, then advice may be sought from a relative/carer/friend acting as a consultee. When reasonable steps have been taken to identify a consultee and one is unavailable, then the researcher must nominate a person to act as in their stead. This person may be involved in the patient's care in a professional capacity but they must have no connection with the research project. A suitable person who might act as a nominated consultee is an independent doctor working with the patient or nominated by the healthcare provider. Consent from the patient will be obtained directly, if they recover promptly, at the earliest opportunity.

11.2.Discontinuation/Withdrawal of Participants from Trial Treatment

11.2.1. Study Withdrawal

We anticipate and have made provision for withdrawal when the emergency exception period is complete; if a patient is assessed and has capacity then they may completely or partially withdraw at any time. This possibility will be made clear as a part of seeking of full written informed consent after the initial emergency procedure. Participants may have the following three options for withdrawal:

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


1) Participants may withdraw from active follow-up and further communication but allow the trial

team to continue to write to their GP and access their medical records and any relevant hospital

data that is recorded as part of routine standard of care; i.e., Radiology/diagnostic test, blood

results and disease progression data etc.

2) Participants can withdraw from the study but permit data obtained up until the point of

with drawal to be retained for use in the study analysis. No further data would be collected after  $\ \ \, = \$ 

withdrawal.

3) Participants can withdraw completely from the study and withdraw the data collected up until

the point of withdrawal. The data already collected would not be used in the final study analysis.

The type of withdrawal and reason for withdrawal will be recorded in the case report form (CRF).

If the participant is withdrawn due to an adverse event, the Investigator will arrange for follow-up visits

or telephone calls until the adverse event has resolved or stabilised.

11.2.2. Participant death

If the participant dies before giving full written consent then we propose to continue using the data

obtained. We would not seek further 'consent' from relatives at the risk of causing undue distress.

11.3.Recruitment

RETRIEVE-AMI is a multi centre study recruiting at the John Radcliffe Hospital and the Newcastle upon

Tyne Hospitals NHS Foundation Trust sites. Participants will be identified as they are being admitted for

primary PCI. They will be approached by a research team member (a primary PCI operator who is also

a member of the clinical care team) who will verbally assent them as explained in section 11.1.1.1. Upon

assent, participant will be randomised to one of the three study arms, by a system based on sealed

Envelope system. Consent will be completed at the post-emergency phase as described in section

11.1.1.3.

11.4. Randomisation

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


Date and version No:22/04/2024 v4.0

Upon assent, participant will be randomised to one of the three study arms, by a system based on sealed envelopes. Randomization will take place in the cathlab once both inclusion and exclusion criteria are verified and assent provided.

11.5. Blinding and code-breaking

Due to the interventional nature of the trial, masking and code-breaking procedures are not applicable.

11.6. Study timeline

Stage 1 – Screening, Assent & Randomisation

Participant identification and assent will proceed as described in sections 10 and 11.1.1.1.1.1.1.2

respectively.

• Diagnostic angiography will be performed in the standard manner using appropriate catheters.

Heparin will be administered as routinely used for PCI. Angiograms will be reviewed to ensure

participation eligibility according to angiographic inclusion/exclusion criteria (section 10.3)

• Once eligibility is confirmed patients will be assented and randomised.

Stage 2 – Baseline assessments

Once the lesion has been crossed with a coronary guidewire, flow will be established with a 1.5mm

semicompliant balloon predilation.

OCT measurements will be performed using a dedicated OCT catheter over the coronary guide wire in

the usual manner for clinical OCT assessment. For Arm 1, the OCT measurements in the baseline

assessment will be treated as the pre-stent measurements as thrombus modification will not be

performed in this group.

Stage 3 – Post-thrombus modification pre-stent assessments

Patients randomised to Arm 2 (thrombus aspiration) or Arm 3 (thrombus retrieval) will undergo the

assessments in this stage.

• Thrombus aspiration (Arm 2) will proceed according to standard clinical practice. In brief, a thrombus

aspiration device (i.e. Export Catheter) will be advanced over the coronary guidewire. Aspiration will

then proceed.

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


• Retrieval thrombectomy (Arm 3) will proceed according to the manufacturer's manual. In brief, a

 $microcatheter \ (e.g.\ Phenom^{TM},\ Marksman^{TM})\ is\ advanced\ over\ the\ guidewire.\ Once\ the\ microcatheter$ 

has traversed the thrombotic occlusion the Solitaire™ X revascularisation device is advanced through

the microcatheter until the usable length of the stent extends past each side of the thrombus in the

vessel. Then the microcatheter is retracted to the proximal radiopaque marker of the stent. As this

retraction occurs the stent self-expands and entangles the thrombus. Next, the microcatheter and

Solitaire  $^{\text{TM}}$  X Revascularisation Device are withdrawn as a unit into the guide catheter under

continuous aspiration (Appendix C).

OCT measurements will be performed using a dedicated OCT catheter over the coronary guide wire in

the usual manner for clinical OCT assessment.

Angiography-derived coronary physiology measurements will be performed with up to two

angiographic views (complementary and separated by an angle of at least 25 degrees) at a frame rate

of 15 frames per second. Maximal hyperaemia will be achieved with an intravenous infusion of

adenosine at a rate of at a rate of 140 mg/kg/min. Since stage 3 is the same as stage 2 for Arm 1

participants, these measurements will be performed at Stage 2.

• Extracted thrombus from aspiration/stent retriever at any stage of the procedure will be collected,

and imaged ex-vivo.

Stage 4 – PCI & post-PCI assessments

PCI will proceed according to clinical practice. Post-dilation will be performed at the operator's

discretion.

OCT measurements will be performed following a successful angiographic PCI result using a dedicated

OCT catheter over the coronary guide wire in the usual manner for clinical OCT assessment.

Angiography-derived coronary physiology measurements will be performed with up to two

angiographic views (complementary and separated by an angle of at least 25 degrees) at a frame rate

Clinical Trial Protocol Template version 15.0


of 15 frames per second. Maximal hyperaemia will be achieved with an intravenous infusion of

adenosine at a rate of at a rate of 140 mg/kg/min.

Stage 5 - Consent & data collection

Patients will be approached for consent according to procedures detailed in section 11.1.1.3. Once consent

has been obtained in-hospital data collection will be completed (section 11.7.1.). ECGs will also be stored.

Stage 6 - 6 month follow-up

At 6 months patients will have a scheduled telephone follow-up to gather relevant clinical information as

detailed in section 11.8.

11.7. Trial Assessments

11.7.1. Data Collection, Patient Reported Outcomes and Clinical Outcomes

Data on the clinical procedures and any devices and/or imaging technologies used will be collected.

Medical history will be taken from the patient once informed consent has been given and relevant sections

of the medical notes and scans may be accessed by the study team. Clinical outcomes and MACCE will be

ascertained at the 6-month telephone follow-up, by accessing relevant sections of the medical records or

by contacting the GP if appropriate.

11.7.2. Optical Coherence Tomography

OCT is a high-resolution intravascular imaging modality that can accurately characterise coronary plaque

morphology and quantify atherothrombotic burden.<sup>4,19</sup> It also has the capability to accurately define the

inner lumen of the native coronary artery allowing to measure the flow area and monitor the structural

integrity of the artery. It is expected therefore to play a key role in identifying target vessel complications

(e.g. dissection, intramural haematoma) and aspects of stent deployment (e.g. stent apposition,

expansion, edge dissection).<sup>20</sup> Finally, OCT has the advantage of having a fast acquisition frame rate and

being relatively inexpensive.

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


11.7.3. Angiography-derived coronary physiology

Coronary physiology measurements during emergency PCI can be used to assess the coronary

microvascular function which is affected amongst other factors by the pre-stenting thrombotic burden and

distal embolisation of atherothrombotic material during angioplasty.3 Indeed, coronary physiology

measurements under adenosine-induced hyperaemia can be employed to characterise microvascular

obstruction and predict the extent of myocardial infarction.<sup>21</sup> Contemporary work enables us to derive

cardiac physiology indices such as quantitative flow ratio non-invasively using coronary angiograms. <sup>22,23</sup>

11.7.4. Extracted Thrombus Imaging

Intracoronary thrombus/plaque material obtained with the use of aspiration/stent-retriever

thrombectomy as part of the procedure will be imaged ex-vivo. Images will be obtained in the

catheterisation laboratory and stored in a pseudonymised format. The extracted thrombus will not be

stored by the study team and will be discarded.

11.7.5. Electrocardiography (ECG)

ECG refers to the measurement of the electrical activity of the heart. It is a routine non-invasive

assessment carried out in patients with suspected or known coronary artery disease.

11.8. Subsequent telephone follow-ups

Participants will have a scheduled telephone follow-up 6 months after their randomisation to the study.

This telephone follow-up will gather information on concurrent medication therapy, patient reported

outcomes, study outcomes and serve as an opportunity to log a participant's recovery progress.

11.9. Definition of End of Trial

Recruitment to the trial will cease as soon as 81 participants have been randomised in the study and have

completed follow-up at 6 months. The trial will end when the last patient exits the study. To ensure that

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


| Date and version No:22/04/2024 v4.0 |
|---|
| the scientific integrity of the trial is maintained, should the target recruitment not be reached by the pre- |
| specified study end-date we will seek an extension of the study |
| specified study end-date we will seek an extension of the study |
| Clinical Trial Protocol Template version 15.0 CONFIDENTIAL |
| © Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019<br> |

#### 12. IDENTIFICATION & DESCRIPTION OF THE INVESTIGATIONAL DEVICE & COMPARATORS

## 12.1. Investigational Device & Comparators

#### 12.1.1. Standalone PCI (Arm 1)

Participants randomised to the standalone PCI arm of the RETRIEVE AMI trial will have standard of care treatment. Participants will undergo PCI with devices and techniques driven by clinical decision making at the patient level and institutional level, and carried out in accordance with local guidelines.

### 12.1.2. Aspiration thrombectomy and PCI (Arm 2)

Participants randomised to Arm 2 of the RETRIEVE AMI trial will have standard of care treatment with manual thrombectomy catheter and PCI. Participants will undergo PCI with devices and techniques driven by clinical decision making at the patient level and institutional level, and carried out in accordance with local guidelines.

## 12.1.3. Investigational arm (Arm 3)

Participants randomised to the stent-retriever thrombectomy arm of the RETRIEVE AMI trial will undergo stent-retriever thrombectomy with the Solitaire™ X Revascularisation Device (Figure 3). The Solitaire™ X revascularisation device has been clinically approved and CE marked for use in acute ischaemic stroke endovascular intervention.¹⁴ Solitaire™ X works by mechanically retrieving the thrombus and restoring blood flow to the area distal to the occlusion. The Solitaire™ X Revascularisation Device is a self-expanding stent designed for dynamic clot integration with radiopaque markers that enhance visualisation of the optimal working length. Features including the range of stent diameters and usable lengths are presented in Appendix B. The device can be used in

Solitaire<sup>TM</sup> X
Revascularization Device

TENYEARS OF INNOVATION

Figure 3: Solitaire<sup>TM</sup> X device

vessels with a diameter between 2.0mm and 5.5mm at the thrombotic occlusion site (Appendix B).

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019 

Commented [FK(O3]: This should be made applicable to both organisations so perhaps"carried out in accordance with the hospital department quideliner."

Commented [RK4R3]: Thank you. Addressed.

**Commented [FK(05]:** This should be made applicable to both organisations so perhaps"carried out in accordance with the hospita department guidelines."

Commented [RK6R5]: Addressed

After a thrombotic occlusion has been identified and crossed with a guidewire, the stent-retriever thrombectomy proceeds as described below (see Appendix C for schematic diagram). A microcatheter (e.g. Phenom<sup>TM</sup>, Marksman<sup>TM</sup>) is advanced over the guidewire. Once the microcatheter has traversed the thrombotic occlusion the Solitaire<sup>TM</sup> X revascularisation device is advanced through the microcatheter until the usable length of the stent extends past each side of the thrombus in the vessel. Then the microcatheter is retracted to the proximal radiopaque marker of the stent. As this retraction occurs the stent self-expands and entangles the thrombus. Finally, the microcatheter and Solitaire<sup>TM</sup> X Revascularisation Device are withdrawn as a unit under continuous aspiration into the guide catheter. PCI will then proceed with devices and techniques driven by clinical decision making at the patient level and institutional level, and carried out in accordance with local guidelines.

12.1.4. Masking (blinding)

Due to the interventional nature of the trial, masking is not applicable.

## 12.1.5. Storage of investigational devices

The Solitaire<sup>™</sup> X Revascularisation Device and Phenom microcatheters will be provided by Medtronic. The OFDI catheters will be provided by Terumo Inc. We will be documenting the number of devices, with their lot numbers, that will be shipped to the John Radcliffe Hospital and Newcastle Upon Tyne Hospitals NHS Foundation Trust. After their delivery, the kit will be stored in designated spaces at both sites and kept in a cool, dry place. We will document on the CRF the LOT number and expiry date for each device for each patient.

#### 12.2. Retriever thrombectomy safety


Stent-retriever thrombectomy is clinically tested and licensed for endovascular intervention in acute ischaemic strokes with large vessel occlusions involving the internal carotid and the first segment of the middle cerebral artery. 14,24 Our proposed pilot in acute coronary syndrome – STEMI patients would therefore represent an off-license application for the Solitaire<sup>TM</sup> X Revascularisation Device. Endovascular intervention for acute ischaemic stroke bears similarities to coronary intervention for acute myocardial Clinical Trial Protocol Template version 15.0 CONFIDENTIAL © Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019

**Commented [FK(07]:** This should be made applicable to both organisations so perhaps"carried out in accordance with the hospita department guidelines."

Commented [RK8R7]: Addressed

infarction. Off license use of retriever thrombectomy in STEMI patients is reported twice in the literature

with no reported complications and a successful recanalization outcome. 15,16

From an anatomical perspective, the Solitaire<sup>TM</sup> X revascularisation device is licensed for interventions in

vessels with a minimum diameter of 2mm and a maximum of 5.5mm depending on the device model used

(see appendix A). The diameter of internal carotid and middle cerebral arteries (arteries for which

Solitaire<sup>™</sup> X intervention is licensed) is reportedly 3.38±1.34mm and 2.45±0.85mm respectively.<sup>25</sup> Our

pilot study is designed to include patients with heart attack due to thrombotic occlusion of a "large caliber"

coronary artery (diameter at the site of occlusion ≥ 3.0 mm). The size range of the target vessel is thus well

within the safety range proposed by the manufacturer (e.g. between 2.0 and 5.5 mm).

From a device perspective, in stroke patients Solitaire™ X revascularisation device failure was reported in

one case (0.8%) in the two pivotal trials that examined this end-point with no significant sequelae.  $^{14,26}$ 

Regarding device related complications in patients randomised to the Solitaire  $^{\text{TM}}$  X revascularisation

device, arterial dissection or perforation was reported in 5/211 (2.3%). Perforations, albeit in the

coronaries are encountered in routine PCI practice in 0.37% of patients<sup>27</sup>, while edge dissections following

stent deployment in 7.7% of patients.<sup>28</sup> The relatively higher perforation with the Solitaire<sup>TM</sup> X device can

be explained by the tortuosity of the intracerebral vessels that are treated as well as the early stage of the

thrombectomy experience in the RCTs and the small sample size. To minimise the potential for coronary

perforations in our trial, we will include patients with thrombotic occlusions involving the right coronary

artery prior to the crux, e.g. in a vessel segment with minimal, if any, tortuosity. Nonetheless, in the event

of a coronary perforation the treatment – angioplasty – is similar to the definitive treatment for the

myocardial infarction.

Finally, stroke in the context of pPCI is reported in 0.25% to 0.5% of STEMI cases<sup>29-31</sup> and in ~0.8% of STEMI

patients with aspiration thrombectomy and PCI.<sup>30</sup> In the Solitaire™ X device trials, the rate of embolisation

to vascular fields proximal to the target vessel is not reported. It is therefore not possible to estimate the

risk of stroke for our trial. However, from a mechanistic perspective stent-retriever thrombectomy is based

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


on the concept of integration of the stent scaffold into the thrombus which in combination with the withdrawal of the stent into the microcatheter and the continuous aspiration on withdrawal renders embolisation of thrombotic material less likely.

# 12.3. Other Interventions

Not applicable

# 13. SAFETY REPORTING

## 13.1. Definitions

| Any untoward medical occurrence, unintended disease or injury or any |
|---|
| untoward clinical signs (including an abnormal laboratory findings) in |
| participants, users or other persons whether or not related to the |
| investigational medical device. This includes events related to the |
| investigational device or comparator, events related to the procedures |
| involved (any procedure in the protocol). For users or other persons |
| this is restricted to events related to the investigational medical device. |
| An adverse event related to the use of an investigational medical device. |
| This definition includes any events resulting from insufficient or |
| inadequate instructions for use, deployment, implantation, installation, |
| or operation, or any malfunction of the investigational device. This |
| definition also includes any event resulting from user error or form |
| intentional misuse of the investigational device. |
| Any untoward medical occurrence that: |
| Results in death |
| Is life-threatening, |
| Requires inpatient hospitalisation or prolongation of existing |
| hospitalisation, |
| Results in persistent or significant disability/incapacity, or |
| Is a congenital anomaly/birth defect. |
| Other important medical events. |

Included herein are device deficiencies that might have led to a serious adverse event if:

- a) suitable action had not been taken or
- b) intervention had not been made or
- c) circumstances had been less fortunate.

These are handled under the SAE reporting system.

Planned hospitalisation for a pre-existing condition, or a procedure required by the trial protocol, without serious deterioration in health, is not considered a serious adverse event.

The term 'life-threatening' in the definition of 'serious' refers to an event in which the patient was at risk of death at the time of the event. It does not refer to an event that hypothetically might have caused death if it were more severe.

Hospitalisation for a pre-existing condition, including elective procedures planned prior to study entry, which has not worsened, does not constitute a serious adverse event.

Other events that may not result in death, are not life threatening, or do not require hospitalisation, may be considered a serious adverse event when, based upon appropriate medical judgement, the event may jeopardise the patient and may require medical or surgical intervention to prevent one of the outcomes listed above.

| Serious Adverse Device | Any untoward medical occurrence that can be attributed wholly or |
|---|---|
| Effect (SADE) | partly to the device, which resulted in any of the characteristics of a |
| | serious adverse event as described above. |
| | Unanticipated Serious Adverse Device Effects (USADE) |
| | Any serious adverse device effect which, by its nature, incidence, |
| | severity or outcome, has not been identified |
| Device deficiency | Inadequacy of a medical device with respect to its identity, quality, |
| | durability, reliability, safety or performance. Device deficiencies include |
| | malfunctions, use errors and inadequate labelling. |
| | Device deficiencies that did not lead to an adverse event, but could have |
| | led to a medical occurrence if suitable action had not been taken, or |
| | intervention had not been made or if circumstances had been less |
| | fortunate |
| User error | Act or omission of an act that results in a different medical device |
| | response than intended by the manufacturer or expected by the user. |
| | Use error includes slips, lapses and mistakes. An unexpected |
| | physiological response of the subject does not itself constitute a use |
| | error. |

## Severity definitions

Mild: awareness of signs or symptoms, that does not interfere with the subject's usual activity or is transient that resolved without treatment and with no sequelae.

Clinical Trial Protocol Template version 15.0


 ${\small \texttt{©} \ Copyright: The \ University \ of \ Oxford \ and \ Oxford \ University \ Hospitals \ NHS \ Foundation \ Trust \ 2019}$ 


Moderate: a sign or symptom, which interferes with the subject's usual activity.

Severe: incapacity with inability to do work or perform usual activities.

Arterial injury classification scheme

Coronary dissections and perforations will be classified according to the established NHLBI and Ellis

classification schemes. 32,33 A significant coronary dissection is defined as a dissection leading to coronary

flow impairment or coronary occlusion.

13.2. Causality

The relationship of each adverse event to the trial device may be determined by the manufacturer and/or

a medically qualified Investigator according to the following definitions:

Not related: The event is clearly related to other factors such as the patients/participants clinical condition,

therapeutic intervention, concomitant medication.

Unlikely: The event is probably produced by other factors such as the patients/participants clinical

condition, therapeutic intervention, concomitant medication and does not follow a known response

pattern to the device

Possibly: The event follows a reasonable temporal relationship form the time of placement/administration

and/or follows a known response pattern to the device but could have been caused by other factors such

as the patients/participants clinical condition, therapeutic intervention, concomitant medication.

Most probable: The event follows a reasonable temporal relationship form the time of

placement/administration and/or follows a known response pattern to the device and could not have been

caused by other factors such as the patients/participants clinical condition, therapeutic intervention,

concomitant medication. Further the event immediately follows the administration/placement of the

device and improves on stopping or removing the device.

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


13.3. Procedures for Recording Adverse Events

All adverse events (including ADEs) and device deficiencies occurring during the course of the study will be

recorded on the CRF whether or not attributed to the trial device. The information recorded will include

but not be limited to:

• A description of the event

The dates of the onset and resolution

Action taken

Outcome

Assessment of relatedness to the device

Whether the AE is serious or not

Whether the AE arises from device deficiency

Whether the AE arises from user error

The severity of events will be assessed on the following scale: 1 = mild, 2 = moderate, 3 = severe.

The CI shall submit to Medtronic a report of AEs and ADEs that occur in Arm 3 of this study. AEs/ADEs

considered related to the device as judged by a medically qualified investigator or the Sponsor will be

followed either until resolution, or the event is considered stable.

It will be left to the Investigator's clinical judgment to decide whether or not an AE/ADE is of sufficient

severity to require the participant's removal from treatment. A participant may also voluntarily withdraw

from treatment due to what he or she perceives as an intolerable AE/ADE. If either of these occurs, the

participant must undergo an end of trial assessment and be given appropriate care under medical

supervision until symptoms cease, or the condition becomes stable.

13.4. Reporting Procedures for Serious Adverse Events

Reporting of all Serious Adverse Events will be done in accordance with the European Commission

Guidelines on Medical Devices Serious Adverse Event Reporting (MEDDEV 2.7/3; December 2010).

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


SAEs/SADEs that pose an immediate risk to patient health or safety will be reported to the trial

TSG/Sponsor immediately or no later than 24 hours after the Investigator is aware and to the device

manufacturer, the MHRA and the REC within 2 calendar days of the Chief Investigator becoming aware of

the event. The SAE form should be emailed to ouhsae.reports@ouh.nhs.uk.

All other reported SAEs/SADEs will be reported to the trial TSG, the Sponsor, device manufacturer and the

MHRA within 7 calendar days of notification, if appropriate. This will not include SAEs that may be expected

as part of the risks of routine care. Adverse device events (SADEs, USADEs) and device deficiencies will also

be reported to the device manufacturer. All SAEs will be followed up to resolution.

SAEs/SADEs will be recorded for a time period starting from verbal assent/investigational device

deployment to 30 days following the use of the device.

#### 13.5. Expectedness

Expectedness will be determined according to the Manufacturers risk analysis report

# 13.6. Trial cessation rules

The trial will be halted early if any of the following occur:

- >2 transient ischaemic attack /ischaemic stroke-related SADEs
- >2 coronary perforation-related SADEs
- > 2 significant coronary dissection-related SADEs

# 13.7. Safety Monitoring Committee – Trial Safety Group (TSG)

The Oxford University Hospitals Trust Trial Safety Group (TSG) will conduct a review of all SAEs/SADEs for the trial reported during the quarter and cumulatively. The aims of this committee include:

- To pick up any trends, such as increases in un/expected events, and take appropriate action
- To seek additional advice or information from investigators where required

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


• To evaluate the risk of the trial continuing and take appropriate action where necessary

# 13.8. Safety of stent-retriever thrombectomy

See Section 12.2.

# 13.9. Safety of intravascular imaging

Intravascular imaging using OCT is often performed during PCI to assist in the procedure. The utilization of this modality typically adds up to 5 minutes to the procedure duration. Use of any intra-coronary device including OCT can cause ischaemia, chest discomfort or, rarely, other local coronary complications during the PCI. However, this is in the context of a PCI procedure where significant interventions such as balloon expansion and stent deployment are already being carried out in the coronary artery, which themselves may cause ischaemia, chest pain that may require the use of analgesia, or other local coronary complications.

#### 14. STATISTICS

#### 14.1. Number of participants

Based on estimates from previously published work<sup>9,34</sup> and our stipulation for inclusion of patients with high thrombotic burden, we anticipate a mean pre-stent thrombus volume of 9.6mm<sup>3</sup> with a standard deviation estimate of 5.1 mm<sup>3</sup> in the standard of care arms. Since this is the first pilot of stent retriever in acute coronary syndromes there is no previous published work that can inform on the expected pre-stent thrombus volume reduction with retriever thrombectomy. We have therefore hypothesised a 33% reduction in mean pre-stent thrombus volume. Using a 1-way pairwise ANOVA with a 2-sided equality, accounting for 2 pairwise comparisons with an  $\alpha$  of 0.05, a sample size of 72 patients would have 80% power to detect a 33% reduction in pre-stent thrombus volume with retriever thrombectomy.<sup>35</sup> The approach that was used accounts for two pairwise comparisons. Indeed, for one such comparison a sample size of n=48 (n=24 for Arm 1 and 24 for Arm 3) would maintain the desired  $\alpha$  of 0.05 and  $\beta$  of 0.2. Given that aspiration thrombectomy was not shown to differ from no thrombus modification, a sample size of n=48 (n=24 for Arm 2 and n=24 for Arm 3) would maintain the desired  $\alpha$  of 0.05 and  $\beta$  of 0.2 for this comparison. The overall sample size is therefore increased by a further n=24 patients for the aspiration thrombectomy group. This leads us to n=72 patients required to show a 33% reduction in pre-stent thrombus burden with a power of 80%. Assuming 12.5% of patients will not have analysable OCT imaging, we plan to enrol 81 patients (n=27 in each group) to ensure the study remains adequately powered.

# 14.2. Analysis of Endpoints

In keeping with our usual practice, we will obtain expert statistical advice from the Centre for Statistics in Medicine (or equivalent) for each specific task. A flow diagram detailing number of participants screened and randomised will be provided. Analysis of the OCT-derived primary and secondary endpoints (including angiography-derived) will be conducted offline in a blinded fashion. Summary statistics, including means, medians, and variances, will be calculated at each time point and for each type of data and group (e.g. baseline characteristics, parameters derived from OCT, angiography-derived coronary physiology). The distribution of the levels will be described. For each parameter an analysis of variance will be carried out.

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


An analysis evaluating for a between group difference in pre-stent thrombus volume will first use an 1-way

ANOVA with a 2-sided equality test to assess for an overall trend. Post-hoc analyses exploring the following

hypotheses i) retriever thrombectomy (Arm 3) is different to no thrombus modification (arm 1) and ii)

retriever thrombectomy (Arm 3) is different to aspiration thrombectomy (Arm 2) will be performed using

the Dunnett test. Control of the Type I error at 5% two-sided significance level due to multiple testing will

be achieved using Dunnett's method.<sup>36</sup> . Missing data for the primary analysis will be dealt with complete

case analysis if data missingness is <10% (<3 cases per group). If missingness is higher, multiple imputation

will be performed instead. Major adverse cardiac and cerebrovascular events will be analysed using

proportions statistical testing (Fisher's exact or  $\chi 2$  tests), yet they represent an exploratory analysis.

14.3. Interim Safety Analysis

Based on the reported coronary perforation (0.37%), coronary dissection (7.7%) and transient ischaemic

attack/ischaemic stroke (0.25-0.8%) rates in contemporary STEMI practice, in a 27-patient arm study, 1

coronary perforation, 1 significant coronary dissection and 1 transient ischaemic attack/ischaemic stroke

may be expected by chance. If >2 (>10%) coronary perforation-related SADEs or >2 significant coronary

dissection-related SADEs or >2 transient ischaemic attack-/ischaemic stroke-related SADEs occur in the

investigational device arm this will be considered too high.

Clinical Trial Protocol Template version 15.0


**15. DATA MANAGEMENT** 

15.1. Source Data

Source documents are where data are first recorded, and from which participants' CRF data are obtained.

These include, but are not limited to, hospital records (from which medical history and previous and

concurrent medication may be summarised into the CRF), ECGs, radiographic and OCT images and

correspondence. Access to relevant source data will be sought for members of the research team.

15.2. Data recording and Record Keeping

The study will comply with the Data Protection Act, which requires data to be anonymised as soon as it is

practical to do so. This will be achieved by assigning participants a unique trial ID number that will be used

in case record forms (CRFs), ECGs, radiographs, OCT and extracted thrombus images (pseudonymisation).

A contact record form linking a participant's unique trial ID number with their personal identifiable data

(name, hospital ID, personal address, emails or telephone numbers) will be used. This form will be kept in

the code break folder, separate from other documents. This form is needed to perform the 6 months

telephone follow-up and to ensure that in case of an emergency participants can be identified and

contacted. The written informed consent form that contains personal data (name and signature) can not

be anonymised, but will be kept in a separate folder to the pseudonymised data and stored securely at the

Oxford University Hospitals NHS Foundation Trust and the Newcastle upon Tyne Hospitals NHS Foundation

Trust.

Study data will be entered into the CRFs by members of the research team after reviewing source data

and/or seeking information from the patient. This data will then be securely stored in an on-site location

with restricted access and will only be accessible by study staff and authorised personnel. Pseudonymised

data from non-Oxford sites can be transferred using appropriately encrypted means to Oxford University

Hospitals NHS Foundation Trust. Source ECG data will be copied, identifiable data will be removed and

subsequently labelled with the trial participant ID number. ECG's will be securely stored alongside the

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


Commented [GS(09]: How will this be done?

Commented [RK10R9]: Hi Steph, we typically use USB/hard drive/email but we don't want to restrict ourselves in the protocol in case of other suitable encrypted ways for data transfer.

participant's CRFs in an on-site location with restricted access and will only be accessible by study staff and

authorised personnel. Radiographic and OCT imaging data will be de-identified using the unique trial

participant ID number before downloading them on to encrypted electronic transfer media and

transferred to be stored on to password protected NHS computers in an on-site location with restricted

access. Pseudonymised data from non-Oxford sites can be transferred using appropriately encrypted

means to Oxford University Hospitals NHS Foundation Trust. In Oxford, extracted thrombus imaging data

will be stored in a de-identified format using the trial participant ID number on to password protected NHS

computers in an on-site location with restricted access.

Personal data (contact record form) will be stored for 12 months after the study has ended, while

pseudonymised research data generated by the study and any research documents with personal

information, such as the consent forms, will be stored for 10 years. All study data and documents will be

stored securely in an on-site location with restricted access. Study data will only be accessed by study staff

and authorised personnel. After analysis is completed, data will be archived in a secure location with

restricted access. After the specified data storage period elapses, the data custodian will agree a date for

destruction and data will be destroyed confidentially at that time.

15.3. Access to Data

Direct access will be granted to authorised representatives from the Sponsor, host institution and the

regulatory authorities to permit trial-related monitoring, audits and inspections.

15.4. Approval to share imaging data with third parties

De-identified research data including imaging data may be shared with the University of Oxford or other

specialised centers in partnership with RETRIEVE-AMI, according to the availability of specialist analysis

techniques that may not be available to the local research team. Data transfer and storage should follow

the processes described in 15.2. Participants will be informed in the information leaflet and sign in the

consent form (if they approve) that their pseudonymised images may in the future be sent to third parties

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


| Date and version No:22/04/2024 v4.0 |
|---|
| for specialist processing. It will be clearly stated that no identifying information will be sent with these |
| imaging data. |
| Clinical Trial Protocol Template version 15.0 CONFIDENTIAL © Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019 |

# **16. QUALITY ASSURANCE PROCEDURES**

# 16.1. Risk assessment

The trial will be conducted in accordance with the current approved protocol, ICH GCP, relevant regulations and standard operating procedures.

# 16.2. Monitoring

Regular monitoring will be performed by the sponsor according to ICH GCP. Data will be evaluated for compliance with the protocol and accuracy in relation to source documents. The monitors will verify that the clinical trial is conducted and data are generated, documented and reported in compliance with the protocol, GCP and the applicable regulatory requirements.

17. PROTOCOL DEVIATIONS

A trial related deviation is a departure from the ethically approved trial protocol or other trial document

or process or from Good Clinical Practice (GCP) or any applicable regulatory requirements. Any deviations

from the protocol will be documented in a protocol deviation form and filed in the trial master file.

All deviations will be reported to the MHRA.

**18. SERIOUS BREACHES** 

A serious breach is defined as "A breach of GCP or the trial protocol which is likely to affect to a significant

degree -

(a) the safety or physical or mental integrity of the subjects of the trial; or

(b) the scientific value of the trial".

In the event that a serious breach is suspected the Sponsor must be contacted within 1 working day. In

collaboration with the C.I., the serious breach will be reviewed by the Sponsor and, if appropriate, the

Sponsor will report it to the REC committee, Regulatory authority and the NHS host organisation within

seven calendar days.

Clinical Trial Protocol Template version 15.0


#### 19. ETHICAL AND REGULATORY CONSIDERATIONS

#### 19.1. Declaration of Helsinki

The Investigator will ensure that this trial is conducted in accordance with the principles of the Declaration of Helsinki.

#### 19.2. Guidelines for Good Clinical Practice

The Investigator will ensure that this trial is conducted in accordance with relevant regulations and with Good Clinical Practice.

#### 19.3. Medical Device Regulations

The Investigator will ensure that this trial is conducted in full conformity with:

- European Commission Medical Device Guidelines relating to the application of the EU Directives
   on Medical Devices
- Guide to European Medical Device Trials and BS EN ISO 14155

# 19.4. Approvals

Following Sponsor approval the protocol, informed consent form and participant information sheet will be submitted to an appropriate Research Ethics Committee (REC), HRA (where required), regulatory authorities (MHRA in the UK), and host institution(s) for written approval.

The Investigator will submit and, where necessary, obtain approval from the above parties for all substantial amendments to the original approved documents.

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


# 19.5. Specific Ethical Considerations for participants in emergency situations

Research in emergency situations is ethically complex because of the urgent nature of the interventions and the often severely compromised capacity of the patient. The processes of enrolment and consent described above, including verbal assent and the involvement of the Advocate represents our attempt to develop a thorough, ethically justified process that both protects patients' rights and interests and enables important research to be done. These processes have been developed in the light of and guided by the provisions laid out in the Mental Capacity Act with special reference to Section 32(9).

# 19.6. Possible risks/discomfort to participants

Patients referred for emergency cardiac catheterization and PCI will undergo this procedure as would routinely be performed. Patients will therefore be informed of the standard of care procedure and its associated risks. All local protocols will be adhered to and only fully trained staff will carry out procedure according to departmental SOPs.

From a research perspective, the PCI procedure time may be lengthened by around 10 minutes to complete the selected study procedures (OCT acquisitions, angiography derived physiology & aspiration/stent retriever thrombectomy). In the context of a PCI procedure that typically lasts approximately 60 minutes. The additional time should not result in any clinically significant difference to the participants. Very occasionally this additional time can result in some back discomfort for patients having to lie on the angiography bed for the additional time period.

Stent-retriever thrombectomy with the Solitaire X revascularisation device is clinically tested and licensed for endovascular intervention in acute ischaemic strokes. Device failure was reported in one case (0.8%) in the two trials that examined this endpoint with no significant sequelae. Device related complications such as arterial dissection or perforation was reported in 5/211 (2.3%) of ischaemic stroke patients randomised to stent-retriever thrombectomy with the Solitaire X revascularisation device. Perforations and edge dissections are encountered in routine PCI practice in 0.37% and 7.7% of patients and interventional cardiologists are familiar with their management. Coronary perforations and significant Clinical Trial Protocol Template version 15.0 CONFIDENTIAL © Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019

dissections are usually treated with a stent which is the treatment these patients will eventually receive

for their heart attack.

Finally, stroke in the context of pPCI is reported in 0.25% to 0.5% of STEMI cases and in  $\sim$ 0.8% of STEMI

patients with aspiration thrombectomy and PCI. In the Solitaire X device trials, the rate of embolisation to

vascular fields proximal to the target vessel is not reported. From a mechanistic perspective, stent-

retriever thrombectomy is based on the concept of integration of the stent scaffold into the thrombus

which in combination with the withdrawal of the stent into the microcatheter and the continuous

aspiration on withdrawal renders embolisation of thrombotic material less likely.

Patients having a heart attack have a higher risk of cardiac mortality, heart failure, periprocedural

myocardial infarction and access-site complications (haematoma, bruising, discomfort) by virtue of the

underlying condition and its treatment with PCI. Additionally, participants who have suffered a heart attack

are frequently re-admitted for a pre-planned procedure to complete revascularisation of their coronary

artery disease. We expect that some combination of these events will be noted in trial participants during

the study follow-up period. Adverse event reporting will proceed as described in section 13.

19.7. Collaboration and Partnership with Commercial Companies & Third parties

The Oxford University Hospitals NHS Foundation Trust (OUHT), the Newcastle upon Tyne Hospitals NHS

Foundation Trust and the RETRIEVE-AMI study receive support from, commercial companies who provide

the devices and technologies related to PCI and other research investigations.

To future proof our study, we may also share research data, including imaging data, with the University of

Oxford or other specialised centres (academic or commercial) in partnership with The Oxford University

Hospitals Trust, the Newcastle upon Tyne Hospitals NHS Foundation Trust and the RETRIEVE-AMI study for

specialist analysis techniques that may not be available to the local research team. We will ensure that

participants are not identifiable from the shared research data.

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


19.8. Feasibility

The Oxford Heart Centre is a state-of-the-art facility which incorporated services in cardiology and cardiac

surgery. The cardiac catheter laboratories are fully equipped to support this study. The Newcastle upon

Tyne Hospitals NHS Foundation Trust is a high volume institution with considerable experience in acute

cardiology research.

19.9. Reporting

The CI shall submit once a year throughout the clinical trial, or on request, an Annual Progress Report to

the REC, the HRA (where required), Medtronic, Terumo Inc, the host organisation, and the Sponsor. A

progress report will also be submitted on a semi-annual basis to Medtronic and Terumo Inc. In addition,

an End of Trial notification and final report will be submitted to the MHRA, the REC, host organisation and

Sponsor. The CI shall make the generated results available to Medtronic and Terumo Inc up to 14 days

before publication or dissemination to the public.

19.10. Participant Confidentiality

The study will comply with the General Data Protection Regulation (GDPR) and Data Protection Act 2018,

which require data to be de-identified as soon as it is practical to do so. The processing of the personal

data of participants will be minimised by making use of a unique participant study number only on all study

documents and any electronic database(s), with the exceptions of i) the contact record and ii) consent

forms. All documents will be stored securely and only accessible by study staff and authorised personnel.

The study staff will safeguard the privacy of participants' personal data. Data management is described in

detail in section 15.

**20. FINANCE AND INSURANCE** 

20.1. Funding

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


RETRIEVE AMI will be supported in kind by Medtronic (Minnesota, US) through the provision of medical

devices and assistance with the MHRA application process. RETRIEVE AMI will also be supported in kind by

Terumo corporation (Tokyo, Japan) through the provision of OFDI (second generation OCT) catheters.

20.2. Insurance

NHS bodies are legally liable for the negligent acts and omissions of their employees. If participants are

harmed whilst taking part in a clinical trial as a result of negligence on the part of a member of the trial

team this liability cover would apply.

Non-negligent harm is not covered by the NHS indemnity scheme. The Oxford University NHS Foundation

Trust, therefore, cannot agree in advance to pay compensation in these circumstances.

In exceptional circumstances an ex-gratia payment may be offered.

21. PUBLICATION POLICY

Data will be owned and supervised by the trust. The Investigators will be involved in reviewing drafts of

the manuscripts, abstracts, press releases and any other publications arising from the study. Authors will

acknowledge that the study was funded by Medtronic and Terumo. Authorship will be determined in

accordance with the ICMJE guidelines and other contributors will be acknowledged. Copies of any

publications connected to this study are available on request from the RETRIEVE-AMI investigators.

22. DEVELOPMENT OF A NEW PRODUCT/ PROCESS OR THE GENERATION OF INTELLECTUAL PROPERTY

Not applicable

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019


#### 23. REFERENCES

- 1. Nowbar AN, Gitto M, Howard JP, Francis DP, Al-Lamee R. Mortality From Ischemic Heart Disease. *Circ Cardiovasc Qual Outcomes* 2019; **12**(6): e005375.
- 2. Braunwald E. The treatment of acute myocardial infarction: the Past, the Present, and the Future. Eur Heart J Acute Cardiovasc Care 2012; 1(1): 9-12.
- 3. Niccoli G, Scalone G, Lerman A, Crea F. Coronary microvascular obstruction in acute myocardial infarction. *Eur Heart J* 2016; **37**(13): 1024-33.
- 4. De Maria GL, Patel N, Wolfrum M, et al. The influence of coronary plaque morphology assessed by optical coherence tomography on final microvascular function after stenting in patients with ST-elevation myocardial infarction. *Coron Artery Dis* 2017; **28**(3): 198-208.
- 5. Vlaar PJ, Svilaas T, van der Horst IC, et al. Cardiac death and reinfarction after 1 year in the Thrombus Aspiration during Percutaneous coronary intervention in Acute myocardial infarction Study (TAPAS): a 1-year follow-up study. *Lancet* 2008; **371**(9628): 1915-20.
- 6. Jolly SS, Cairns JA, Yusuf S, et al. Outcomes after thrombus aspiration for ST elevation myocardial infarction: 1-year follow-up of the prospective randomised TOTAL trial. *Lancet* 2016; **387**(10014): 127-35.
- 7. Lagerqvist B, Fröbert O, Olivecrona GK, et al. Outcomes 1 Year after Thrombus Aspiration for Myocardial Infarction. *New England Journal of Medicine* 2014; **371**(12): 1111-20.
- 8. Higuma T, Soeda T, Yamada M, et al. Does Residual Thrombus After Aspiration Thrombectomy Affect the Outcome of Primary PCI in Patients With ST-Segment Elevation Myocardial Infarction?: An Optical Coherence Tomography Study. *JACC: Cardiovascular Interventions* 2016; **9**(19): 2002-11.
- 9. Bhindi R, Kajander OA, Jolly SS, et al. Culprit lesion thrombus burden after manual thrombectomy or percutaneous coronary intervention-alone in ST-segment elevation myocardial infarction: the optical coherence tomography sub-study of the TOTAL (ThrOmbecTomy versus PCI ALone) trial. *Eur Heart J* 2015; **36**(29): 1892-900.
- 10. Berkhemer OA, Fransen PSS, Beumer D, et al. A Randomized Trial of Intraarterial Treatment for Acute Ischemic Stroke. *New England Journal of Medicine* 2014; **372**(1): 11-20.
- 11. Goyal M, Demchuk AM, Menon BK, et al. Randomized Assessment of Rapid Endovascular Treatment of Ischemic Stroke. *New England Journal of Medicine* 2015; **372**(11): 1019-30.
- 12. Campbell BCV, Mitchell PJ, Kleinig TJ, et al. Endovascular Therapy for Ischemic Stroke with Perfusion-Imaging Selection. *New England Journal of Medicine* 2015; **372**(11): 1009-18.
- 13. Jovin TG, Chamorro A, Cobo E, et al. Thrombectomy within 8 Hours after Symptom Onset in Ischemic Stroke. *New England Journal of Medicine* 2015; **372**(24): 2296-306.
- 14. Saver JL, Goyal M, Bonafe A, et al. Stent-retriever thrombectomy after intravenous t-PA vs. t-PA alone in stroke. *N Engl J Med* 2015; **372**(24): 2285-95.

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019

- 15. Bhoopalan K, Rajendran R, Alagarsamy S, Kesavamoorthy N. Successful extraction of refractory thrombus from an ectatic coronary artery using stent retriever during primary angioplasty for acute myocardial infarction: a case report. *European Heart Journal Case Reports* 2019; **3**(1).
- 16. Patel N, Badiye A, Yavagal DR, Mendoza CE. Stent-Based Mechanical Thrombectomy in Left Main Coronary Artery Thrombus Presenting as ST-Segment Elevation Myocardial Infarction. *JACC: Cardiovascular Interventions* 2017; **10**(3): 302.
- 17. Alessandro S, Angelo Q, Marco C, et al. A prospective, first-in-human use of the NeVa mechanical thrombectomy device for patients with acute coronary syndromes. *EuroIntervention* 2022.
- 18. Jakob M, Spasojevic D, Krogmann ON, Wiher H, Hug R, Hess OM. Tortuosity of coronary arteries in chronic pressure and volume overload. *Catheterization and Cardiovascular Diagnosis* 1996; **38**(1): 25-31.
- 19. Kajander OA, Koistinen LS, Eskola M, et al. Feasibility and repeatability of optical coherence tomography measurements of pre-stent thrombus burden in patients with STEMI treated with primary PCI. *Eur Heart J Cardiovasc Imaging* 2015; **16**(1): 96-107.
- 20. Ali ZA, Karimi Galougahi K, Maehara A, et al. Intracoronary Optical Coherence Tomography 2018: Current Status and Future Directions. *JACC Cardiovasc Interv* 2017; **10**(24): 2473-87.
- 21. De Maria GL, Alkhalil M, Wolfrum M, et al. Index of Microcirculatory Resistance as a Tool to Characterize Microvascular Obstruction and to Predict Infarct Size Regression in Patients With STEMI Undergoing Primary PCI. *JACC Cardiovasc Imaging* 2019; **12**(5): 837-48.
- 22. Tu S, Barbato E, Köszegi Z, et al. Fractional Flow Reserve Calculation From 3-Dimensional Quantitative Coronary Angiography and TIMI Frame Count: A Fast Computer Model to Quantify the Functional Significance of Moderately Obstructed Coronary Arteries. *JACC: Cardiovascular Interventions* 2014; **7**(7): 768-77.
- 23. Tu S, Xu L, Lightart J, et al. In vivo comparison of arterial lumen dimensions assessed by coregistered three-dimensional (3D) quantitative coronary angiography, intravascular ultrasound and optical coherence tomography. *Int J Cardiovasc Imaging* 2012; **28**(6): 1315-27.
- 24. Albers GW, Marks MP, Kemp S, et al. Thrombectomy for Stroke at 6 to 16 Hours with Selection by Perfusion Imaging. *New England Journal of Medicine* 2018; **378**(8): 708-18.
- 25. Tarasow E, Abdulwahed Saleh Ali A, Lewszuk A, Walecki J. Measurements of the middle cerebral artery in digital subtraction angiography and MR angiography. *Med Sci Monit* 2007; **13 Suppl 1**: 65-72.
- 26. Saver JL, Jahan R, Levy El, et al. Solitaire flow restoration device versus the Merci Retriever in patients with acute ischaemic stroke (SWIFT): a randomised, parallel-group, non-inferiority trial. *The Lancet* 2012: **380**(9849): 1241-9
- 27. Kinnaird T, Kwok CS, Davies R, et al. Coronary perforation complicating percutaneous coronary intervention in patients presenting with an acute coronary syndrome: An analysis of 1013 perforation cases from the British Cardiovascular Intervention Society database. *Int J Cardiol* 2020; **299**: 37-42.

Clinical Trial Protocol Template version 15.0


© Copyright: The University of Oxford and Oxford University Hospitals NHS Foundation Trust 2019

- 28. Kobayashi N, Mintz GS, Witzenbichler B, et al. Prevalence, Features, and Prognostic Importance of Edge Dissection After Drug-Eluting Stent Implantation: An ADAPT-DES Intravascular Ultrasound Substudy. *Circ Cardiovasc Interv* 2016; **9**(7): e003553.
- 29. Myint PK, Kwok CS, Roffe C, et al. Determinants and Outcomes of Stroke Following Percutaneous Coronary Intervention by Indication. *Stroke* 2016; **47**(6): 1500-7.
- 30. Jolly SS, James S, Dzavik V, et al. Thrombus Aspiration in ST-Segment-Elevation Myocardial Infarction: An Individual Patient Meta-Analysis: Thrombectomy Trialists Collaboration. *Circulation* 2017; **135**(2): 143-52.
- 31. Shoji S, Kohsaka S, Kumamaru H, et al. Stroke After Percutaneous Coronary Intervention in the Era of Transradial Intervention. *Circulation: Cardiovascular Interventions* 2018; **11**(12): e006761.
- 32. Bittl JA, Ryan TJ, Jr., Keaney JF, Jr., et al. Coronary artery perforation during excimer laser coronary angioplasty. The percutaneous Excimer Laser Coronary Angioplasty Registry. *J Am Coll Cardiol* 1993; **21**(5): 1158-65.
- 33. Ellis SG, Ajluni S, Arnold AZ, et al. Increased coronary perforation in the new device era. Incidence, classification, management, and outcome. *Circulation* 1994; **90**(6): 2725-30.
- 34. Amabile N, Hammas S, Fradi S, et al. Intra-coronary thrombus evolution during acute coronary syndrome: regression assessment by serial optical coherence tomography analyses. *European Heart Journal Cardiovascular Imaging* 2014; **16**(4): 433-40.
- 35. Chow S-C, Shao J, Wang H, Lokhnygina Y. Sample size calculations in clinical research: chapman and hall/CRC; 2017.
- 36. Dunnett CW. A Multiple Comparison Procedure for Comparing Several Treatments with a Control. Journal of the American Statistical Association 1955; **50**(272): 1096-121.

# 24. APPENDIX A: Trial flow chart



# 25. APPENDIX B: Vessel reference diameters for device sizing

| Model | Recommended<br>Vessel<br>Diameter <sup>A</sup><br>(mm) | | Minimum<br>Microcatheter<br>ID<br>(inch) | | Push Wire<br>Length | Stent<br>Diameter | Usable<br>Length <sup>B</sup> | Stent<br>Length | Length from<br>Distal Tip to<br>Flourosafe<br>Marker | Radiopaque<br>Markers | | Radiopaque<br>Stent Markers<br>Spacing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (min) | (max) | (min) | (max) | (cm) | (mm) | (mm) | (mm) | (cm) | Distal | Prox. | (mm) |
| SFR4-4-20-05 | 2.0 | 4.0 | 0.021 | 0.027 | 200 | 4.0 | 20.0 | 31.0 | <130 | 3 | 1 | 5 |
| SFR4-4-20-10 | 2.0 | 4.0 | 0.021 | 0.027 | 200 | 4.0 | 20.0 | 31.0 | <130 | 3 | 1 | 10 |
| SFR4-4-40-10 | 2.0 | 4.0 | 0.021 | 0.027 | 200 | 4.0 | 40.0 | 50.0 | <130 | 3 | 1 | 10 |
| SFR4-6-20-10 | 2.0 | 5.5 | 0.021 | 0.027 | 200 | 6.0 | 20.0 | 31.0 | <130 | 4 | 1 | 10 |
| SFR4-6-24-06 | 2.0 | 5.5 | 0.021 | 0.027 | 200 | 6.0 | 24.0 | 37.0 | <130 | 4 | 1 | 6 |
| SFR4-6-40-10 | 2.0 | 5.5 | 0.021 | 0.027 | 200 | 6.0 | 40.0 | 47.0 | <130 | 4 | 1 | 10 |

A. Based on the smallest vessel diameter at thrombus site.

Up to 3 retrieval passes<sup>a</sup>

I. TRAVI 15188 Rev. A. Z. TRAVI 1593 Rev. A. 3. Compared to Solitare "Platnum. A. 71042-001 Rev. B. Umansky, F. et al. Microsurgical anatomy of the proximal segments of the mode cerebral astery. 6. TRAVI 1503 Rev. A. 7. TRAVI 2180 Rev. A. B. DWSSFG 13XXXVVVyy-22 Rev. B. 9. DWSSFG 13XXVVVyy-22 Rev. B. 9. DWSSFG 13XXVVVyy-22 Rev. B. 9. DWSSFG 13XXVVVyy-22 Rev. B. 9. DWSSFG 13XXVVVyy-22 Rev. B. 9. DWSSFG 13XXVVVYy-22 Rev. B. 9. DWSSFG 13XXVVVYy-22 Rev. B. 9. DWSSFG 13XXVVVYy-22 Rev. B. 9. DWSSFG 13XXVVVYY-22 Rev. B. 9. DWSSFG 13XXVVVYY-22 Rev. B. 9. DWSSFG 13XXVVYY-22 Rev. B. 9. DWSSFG 13XXVYY-22 Rev. B. 9. DWSSFG 13XXVXYY-22 Rev. B. 9. DWSSFG 13XXVXXYY-22 Rev. B. 9. DWSSFG 13XXVXXYY-22 Rev. B. 9. DWSSFG 13XXVXXYY-22 REV. B. 9. DWSSFG 13XXVXXYY-22 REV. B. 9. DWSSFG 13XXVXXXXXXXXXXXXX

# 26. APPENDIX C: Schematic diagram of device operation



Figure 4 Line diagram to illustrate the technique of using the thrombus retrieval device. (A) The vessel with thrombus is crossed with a workhorse wire that was pre-loaded with a Rebar micro-catheter. (B) Rebar micro-catheter was advanced beyond the thrombus. (C) The wire was removed; an appropriate sized Solitaire AB device was back loaded and advanced to the tip of the micro-catheter positioned beyond the thrombus. (D) The micro-catheter was pulled back maintaining the tip of the device at the same position. This makes the stent expand and trap the thrombus between its struts. (E) The stent device is then pulled back into the micro-catheter along with the trapped thrombus. (F) Once the device is completely within the micro-catheter the whole system is pulled out.

Schematic diagram of device operation<sup>15</sup>

# 27. APPENDIX D: Amendment history

| Amendment<br>No. | Protocol<br>Version No. | Date issued | Author(s) of changes | Details of Changes made |
|---|---|---|---|---|
| 1 | V1.3 | 21/01/2022 | Rafail A Kotronias<br>Giovanni L De<br>Maria | Sample size increase |
| 2 | V2 | 21/12/2022 | Rafail A Kotronias<br>Giovanni L De<br>Maria | Changes in inclusion and exclusion criteria |
| 3 | v3.0 | 02/10/2023 | Rafail A Kotronias<br>Giovanni L De<br>Maria | Inclusion of an additional site Extension of recruitment period |